CLINICAL TRIAL: NCT01866644
Title: Effectiveness of N-acetylcysteine on Preservation Solution During Liver Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NAC400
Record Dates: First submitted 2012-04-18; First posted 2013-05-31 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-06

CONDITIONS: Unspecified Complication of Liver Transplant
Keywords: Liver transplantation, n-acetylcysteine
MeSH Terms: interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Experimental): At portal level, a cannula is inserted with the usual technique of infusion of 3000 ml of preservation fluid to free fall as containing or not scrambling inserted by the NAC scrub nurse then (400 mg of N-acetylcysteine at 10%, 4 ml ).
  Interventions: Drug: N-acetylcysteine
- Saline (Placebo Comparator): With usual technique
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: N-acetylcysteine — Bath transplanted liver with N-acetylcysteine
  Other Names: Flumil Solution injectable 300 Mg
  Arms: N-acetylcysteine
Drug: Saline — Bath saline transplanted liver
  Other Names: It's not describe in a protocol
  Arms: Saline

SUMMARY:
Evaluate the effectiveness of the administration produced antioxidant N-acetylcysteine (NAC), decreasing the incidence of primary graft dysfunction and primary failure. The degree of dysfunction will be monitored by the method of LIMON, metabonomics techniques and according to the latest published validation Liver Transplantation (16 943-949 2010), total billirrubina greater than 10 mg / dl, INR greater than 1.6 in the seventh postoperative day and alanine or aspartate aminotransferase greater than 2000 IU / L in the first seven days. Liver dysfunction is considered, the presence of a transaminase value> 2000 IU / L 1-7 postoperative day or BT> 10 mg / dl or INR> 1.6, both only in the 7th postoperative day (Olthoff et al Liver Transplantation 16,943 -949 2010).

DETAILED DESCRIPTION:
The reason of this study is to evaluate the efficacy of the use of n-acetylcysteine in liver transplant, by administering it in the perfusion liquid, at the time of extraction of the liver of the donor to improve the damage caused by ischemia / reperfusion. The dose is 400 mg in the portal perfusion liquid.

The study included all considered valid and perfused livers. Patients are randomized to contain no drug or n-acetylcysteine by randomization. Then analyzed using blood tests and in the receiver and daily during the first seven days post-transplant hepatic dysfunction parameters, in order to objectify if liver function improves after administration of the antioxidant (n-acetylcysteine ). Safety assessments were performed with intraoperative monitoring anesthetic depth, postoperative parameters of liver and kidney function and graft pathologic examination after perfusion.

ELIGIBILITY:
Inclusion Criteria:

* All grafts perfused by extraction for liver transplantation.

Exclusion Criteria:

* < 18 years
* Allergy to NAC
* Grafts considered invalid for liver transplantation after perfusion
* Hepatitis fulminant
* Retransplantation
* Split
* > 10 hours of cold ischemia
* Patients with asthma

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The incidence of primary graft dysfunction and primary failure | One week after treatment
  Evaluate the incidence of primary graft dysfunction and primary failure in each group of treatment.

SECONDARY OUTCOMES:
To assess the existence of side effects from the use of n-acetylcysteine on liver preservation solution usual. | One week after treatment
Reduction of postoperative renal disfunction | One week after treatment
Assess levels of glutathione stores achieved following administration of NAC | During harvesting
  During the harvesting and implantation in the recipient liver three liver biopsies will be performed which will be assessed by determining metabonomics metabolites of the transsulfuration pathway and GSH levels.
Histological changes | During harvesting
  Two biopsies which are going to be done in donor graft before and after reperfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Lopez Andujar, PhD, Principal Investigator — Hospital Universitario La Fe; Concepcion Gómez i Gavara, MD, Study Chair — Hospital Universitario La Fe
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Spain

REFERENCES:
- [Background] Zafarullah M, Li WQ, Sylvester J, Ahmad M. Molecular mechanisms of N-acetylcysteine actions. Cell Mol Life Sci. 2003 Jan;60(1):6-20. doi: 10.1007/s000180300001. PMID 12613655
- [Background] De Rosa SC, Zaretsky MD, Dubs JG, Roederer M, Anderson M, Green A, Mitra D, Watanabe N, Nakamura H, Tjioe I, Deresinski SC, Moore WA, Ela SW, Parks D, Herzenberg LA, Herzenberg LA. N-acetylcysteine replenishes glutathione in HIV infection. Eur J Clin Invest. 2000 Oct;30(10):915-29. doi: 10.1046/j.1365-2362.2000.00736.x. PMID 11029607
- [Background] Abstracts of the Brain Research Association meeting, Mechanisms of Recovery of Function after Brain Damage. Oxford, U.K., 11 January 1988. Neurosci Lett Suppl. 1988;32:S107-17. No abstract available. PMID 2897100
- [Background] Himmelfarb J, Hakim RM. Oxidative stress in uremia. Curr Opin Nephrol Hypertens. 2003 Nov;12(6):593-8. doi: 10.1097/00041552-200311000-00004. PMID 14564195
- [Background] Molnar Z, Szakmany T, Koszegi T. Prophylactic N-acetylcysteine decreases serum CRP but not PCT levels and microalbuminuria following major abdominal surgery. A prospective, randomised, double-blinded, placebo-controlled clinical trial. Intensive Care Med. 2003 May;29(5):749-55. doi: 10.1007/s00134-003-1723-1. Epub 2003 Apr 8. PMID 12682719
- [Background] Taniyama Y, Griendling KK. Reactive oxygen species in the vasculature: molecular and cellular mechanisms. Hypertension. 2003 Dec;42(6):1075-81. doi: 10.1161/01.HYP.0000100443.09293.4F. Epub 2003 Oct 27. PMID 14581295
- [Background] Raj DS, Lim G, Levi M, Qualls C, Jain SK. Advanced glycation end products and oxidative stress are increased in chronic allograft nephropathy. Am J Kidney Dis. 2004 Jan;43(1):154-60. doi: 10.1053/j.ajkd.2003.09.021. PMID 14712439
- [Background] Rank N, Michel C, Haertel C, Lenhart A, Welte M, Meier-Hellmann A, Spies C. N-acetylcysteine increases liver blood flow and improves liver function in septic shock patients: results of a prospective, randomized, double-blind study. Crit Care Med. 2000 Dec;28(12):3799-807. doi: 10.1097/00003246-200012000-00006. PMID 11153617
- [Background] Taut FJ, Schmidt H, Zapletal CM, Thies JC, Grube C, Motsch J, Klar E, Martin E. N-acetylcysteine induces shedding of selectins from liver and intestine during orthotopic liver transplantation. Clin Exp Immunol. 2001 May;124(2):337-41. doi: 10.1046/j.1365-2249.2001.01531.x. PMID 11422213
- [Background] Thies JC, Teklote J, Clauer U, Tox U, Klar E, Hofmann WJ, Herfarth C, Otto G. The efficacy of N-acetylcysteine as a hepatoprotective agent in liver transplantation. Transpl Int. 1998;11 Suppl 1:S390-2. doi: 10.1007/s001470050505. PMID 9665023
- [Background] Marczin N, Bundy RE, Hoare GS, Yacoub M. Redox regulation following cardiac ischemia and reperfusion. Coron Artery Dis. 2003 Apr;14(2):123-33. doi: 10.1097/00019501-200304000-00005. No abstract available. PMID 12655276
- [Background] Selzner N, Rudiger H, Graf R, Clavien PA. Protective strategies against ischemic injury of the liver. Gastroenterology. 2003 Sep;125(3):917-36. doi: 10.1016/s0016-5085(03)01048-5. PMID 12949736
- [Background] D'Amico F, Vitale A, Gringeri E, Valmasoni M, Carraro A, Brolese A, Zanus G, Boccagni P, D'Amico DF, Cillo U. Liver transplantation using suboptimal grafts: impact of donor harvesting technique. Liver Transpl. 2007 Oct;13(10):1444-50. doi: 10.1002/lt.21268. PMID 17902131
- [Background] Lopez-Andujar R, Deusa S, Montalva E, San Juan F, Moya A, Pareja E, DeJuan M, Berenguer M, Prieto M, Mir J. Comparative prospective study of two liver graft preservation solutions: University of Wisconsin and Celsior. Liver Transpl. 2009 Dec;15(12):1709-17. doi: 10.1002/lt.21945. PMID 19938119
- [Background] Pedotti P, Cardillo M, Rigotti P, Gerunda G, Merenda R, Cillo U, Zanus G, Baccarani U, Berardinelli ML, Boschiero L, Caccamo L, Calconi G, Chiaramonte S, Dal Canton A, De Carlis L, Di Carlo V, Donati D, Montanaro D, Pulvirenti A, Remuzzi G, Sandrini S, Valente U, Scalamogna M. A comparative prospective study of two available solutions for kidney and liver preservation. Transplantation. 2004 May 27;77(10):1540-5. doi: 10.1097/01.tp.0000132278.00441.cf. PMID 15239618
- [Background] Varadarajan R, Golden-Mason L, Young L, McLoughlin P, Nolan N, McEntee G, Traynor O, Geoghegan J, Hegarty JE, O'Farrelly C. Nitric oxide in early ischaemia reperfusion injury during human orthotopic liver transplantation. Transplantation. 2004 Jul 27;78(2):250-6. doi: 10.1097/01.tp.0000128188.45553.8c. PMID 15280686
- [Derived] Gomez-Gavara C, Moya-Herraiz A, Hervas D, Perez-Rojas J, LaHoz A, Lopez-Andujar R. The Potential Role of Efficacy and Safety Evaluation of N-Acetylcysteine Administration During Liver Procurement. The NAC-400 Single Center Randomized Controlled Trial. Transplantation. 2021 Oct 1;105(10):2245-2254. doi: 10.1097/TP.0000000000003487. PMID 33044432